CLINICAL TRIAL: NCT00492817
Title: Phase I/II Evaluation of Single Session Stereotactic Body Radiotherapy for Spinal or Paraspinal Metastases
Brief Title: Evaluation of Single Session Stereotactic Body Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0445; NCI-2012-01499 (Registry Identifier: NCI CTRP- Clinical Trials Reporting Registry)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Spinal Neoplasms
Keywords: Spinal Neoplasms; Paraspinal Metastases; Stereotactic Body Radiotherapy; CT-on-Rails; Spinal Cord; SBRT
MeSH Terms: conditions — Spinal Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Single Session Stereotactic Body Radiotherapy (SBRT) (Experimental): On day 1 of radiation treatment, a CT scan using CT-on-Rails in the same treatment room, immediately before the radiation treatment will be performed.
  Interventions: Procedure: Stereotactic Body Radiotherapy

INTERVENTIONS:
Procedure: Stereotactic Body Radiotherapy — On day 1 of radiation treatment, a CT scan using CT-on-Rails in the same treatment room, immediately before the radiation treatment will be performed.
  Other Names: SBRT

SUMMARY:
The goal of this clinical research study is to find out if stereotactic body radiotherapy to the spine using computerized tomography (CT)-on-Rails is safe and effective in the treatment of metastatic spine tumors.

Objectives:

* Establish the safety and efficacy of using stereotactic body radiotherapy (SBRT) to treat spine and para-spinal tumors in a single session.
* Document frequency and severity of pain, symptoms and symptom interference, as well as quality of life before and after treatment.
* Document changes in neurological function at defined intervals compared to pre-treatment neurological function.

DETAILED DESCRIPTION:
CT-on-Rails is a system that places the radiation treatment machine in the same room as the CT scanner so that the CT scanner can help deliver radiation more precisely.

You will have a MRI of the spine within 1 month before registration on this study. You will also fill out a health survey, a symptom inventory, and a Brief Pain Inventory within 1 week before registration. Each of these surveys should take about 5 minutes to complete. You will have a CT-simulation. The simulation is like a CT scan where a special body frame is used to keep you from moving during scanning and later radiation treatment. However, no radiation is delivered during the simulation. You will be asked questions about your medical history and have a complete neurological exam during your first consultation, before registration. The neurological exam involves testing upper and lower motor strength, sensation to light touch, reflexes, a mental exam, and an evaluation of the way you walk.

Radiation treatment will last between 2 and 2 1/2 hours and will be given on 1 day about 1 to 1 1/2 weeks after you had the simulation. You will have a device (similar to plastic wrap) placed around you that will hold you still during the treatment. You will be checked for level of pain and/or discomfort before starting each session of radiation, and you may take pain medications before starting each session. All participants will be treated with radiation therapy that is guided by the CT-on-Rails procedure. On the day of radiation, you will also receive a CT scan using CT-on-Rails in the same treatment room, immediately before the radiation treatment.

During treatment, a physician will be monitoring you for any side effects. If you experience severe side effects, radiation treatment will be stopped, and you will be taken off study. After treatment on this study ends, you will have telephone, mail, or facsimile (Fax) follow-ups scheduled at 1, 2, 3, 4, and 8 weeks after radiation. You will be asked questions about any side effects or pain you are experiencing and any other therapies you may have started.

You will have follow-up visits scheduled at 3, 6, 9, 12, 18, and 24 months and then every 6 months for the rest of your life. At all follow-up visits, you will be asked questions about your medical history, have a neurological exam, and your neurologic function will be evaluated. Any pain medication you are taking will be noted. You will be asked to have a MRI of the spine at 3, 6, 9, 12,18, and 24 months, then once a year for the rest of your life. You will also be asked to complete 3 questionnaires to evaluate your symptoms, pain, and quality of life at each follow-up visit. Each questionnaire should take around 5 minutes to complete.

This is an investigational study. The equipment used in this study are FDA-approved medical devices and are commercially available. However, the way the devices are being used in this study is experimental. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographically documented spine or paraspinal metastasis demonstrated on spine MRI within 4 weeks of registration
2. Maximum of 2 metastatic sites in the spine to be irradiated in single session
3. Informed consent for irradiation of spinal or para-spinal tumor (s)
4. Diagnosis of cancer including but not limited to lung (non-small cell and small cell), breast, prostate, renal cell, melanoma, gastrointestinal, and germ cell tumors, unknown primary tumors
5. Karnofsky performance status of at least 40 (ie not requiring active hospitalization)

Exclusion Criteria:

1. Worsening neurological status due to radiographic evidence of spinal cord compression requiring immediate surgical decompression or emergent conventional external radiation therapy.
2. Delay in initiation of radiation treatment would be potentially detrimental to neurological outcome
3. Prior irradiation to current site of interest in the spine
4. Spinal metastasis in the cervical spine are not eligible for treatment
5. Unstable spine requiring surgical stabilization.
6. Sites outside the spine (eg. lung, liver) are not eligible for treatment
7. Patients currently receiving, or who have received chemotherapy within 30 days are not eligible
8. Inability to tolerate lying flat on treatment couch for greater than 30 minutes.
9. Patient with multiple myeloma
10. Patients unable to undergo MRI of the spine
11. Patients with pacemakers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-10-13 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 64
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Complete Pain Relief Using Stereotactic Body Radiotherapy (SBRT) to Treat Spine and Para- Spinal Tumors in a Single Session
Description: To measure 6-month complete pain relief, i.e., 6-month "pain worst" from the BPI being zero
Time Frame: Six months after completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 61
Participants | 18

2. Primary Outcome: Local Tumor Control Rate
Description: Local tumor control rate as measured based on spinal MRI showing absence of progression
Time Frame: local tumor control rate, the time frame is up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 61
Participants | 48

3. Primary Outcome: Paralysis (Grade 4 Motor Neuropathy)
Description: Evidence of paralysis (Grade 4 motor neuropathy) casued by radiation myelitis
Time Frame: Up to 24 months after radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 61
Participants | 0

ADVERSE EVENTS:
Time Frame: Approximately 1 year, 9 months
Arm/Group | Single Session Stereotactic Body Radiotherapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 63/71
Serious Adverse Events (participants affected / at risk) | 7/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Session Stereotactic Body Radiotherapy (SBRT) (N=71)
Nephrostomy tube placement, Malfunctioning prostomy (Renal and urinary disorders) | 1
Esophageal stricture (Gastrointestinal disorders) | 2
Hemorrhage (Blood and lymphatic system disorders) | 1
Diarrhea (General disorders) | 2
Neroforaminal stenosis and nerve root compression (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT00492817/Prot_SAP_000.pdf